CLINICAL TRIAL: NCT03502629
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of GB226 for the Treatment of Chinese Population With Relapsed and Refractory Peripheral T Cell Lymphoma (PTCL)
Brief Title: Clinical Trial in Chinese Patients of Relapsed and Refractory Peripheral T Cell Lymphoma (GB226)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gxplore-002
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB226 3mg/kg every 2 weeks (Experimental): Geptanolimab Injection, 3mg/kg every 2 weeks
  Interventions: Biological: GB226

INTERVENTIONS:
Biological: GB226 — 3mg/kg treat every 2 weeks
  Other Names: Recombinant humanized anti-PD-1 monoclonal antibody injection; Geptanolimab

SUMMARY:
It is a multi-center, prospective, open-label, two-stage optimized design, single-arm, phase II clinical study to evaluate the efficacy and safety of GB226 for the treatment of relapsed and refractory peripheral T cell lymphoma (PTCL), and to evaluate the immunogenicity of GB226.

DETAILED DESCRIPTION:
GB226, 3mg/kg/time, is intravenously infused once every two weeks until disease progression, intolerable toxicity or study withdrawal decided by the investigator/subject.

It is expected that each subject will be followed for 2 years. Subjects receiving GB226 treatment will be followed once every 2 weeks to the end of this study. If the patients terminate the treatment and their imaging assessment shows no progressive disease (PD), they should be followed once every 6 weeks until progressive disease (imaging evaluation). If the patients have progressive disease (imaging assessment), they should be followed every 3 months until the end of this study or premature withdrawal from the study. Relevant tests and evaluation should be completed at each visit according to standard of care. The follow-up visits can be performed by telephone.

During the study, subjects must complete one imaging test and efficacy evaluation every 6 weeks until disease progression. Moreover, patients should be closely monitored for adverse events from subject enrollment to 30 days after the last dosing

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older, male or female;
2. Understand study procedures and contents, and voluntarily sign the written informed consent form;
3. Histologically confirmed relapsed or refractory PTCL patients who had received systemic treatment at least once but had failed to or cannot tolerate the treatment, and/or who cannot be treated with effective standard therapies currently.
4. Available to provide tissue sample for pathological diagnosis;
5. ECOG score of 0-1;
6. Life expectancy≥3 months;
7. Computed tomography (ct) scans performed within 28 days of study administration should show the presence of at least one of two vertical orientationsThe tumor lesions that could be measured were defined, with the longest diameter of intranode lesion > 1.5cm and the longest diameter of extranode lesion > 1.0cm (according to2014 lugano standard)
8. Systemic chemotherapy, systemic or local palliative radiotherapy, target therapy has been completed for at least 4 weeks before enrollment.
9. Systemic corticosteroids (prednisone > 10 mg/day or equivalent dose) has been discontinued at least 2 weeks before enrollment;
10. Autologous hematopoietic stem cell transplantation (ASCT) has been completed at least 4 weeks before enrollment;
11. Before enrollment, major surgery requiring general anesthesia must have been completed at least 4 weeks; surgery requiring local anesthesia/epidural anesthesia must have been completed at least 2 weeks and the patients have recovered; skin biopsy requiring local anesthesia has been completed at least 1 hour.
12. The previous anti-tumor biotherapy (tumor vaccine aimed at controlling tumor, cytokine or growth factor) has been completed at least 4 weeks before enrollment.
13. For routine blood tests: hemoglobin ≥ 80 g/L, neutrophil ≥ 1.0 ×109/L, platelet ≥ 80×109/L;
14. Serum creatinine ≤ 1.5×ULN or creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula);
15. Total bilirubin < 1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times the upper limit of normal (ULN);
16. Thyroid function indicators: thyroid-stimulating hormone (TSH) and free thyroxine (FT3/FT4) are within the normal range;
17. The adverse reactions caused by the previous treatment should recover to grade 1 and below (except alopecia);
18. Females of child-bearing potential have negative serum pregnancy test; males or females agree to adopt medically confirmed contraceptive measures during the entire study and within 6 months after the end of this study.
19. Patients can receive follow-up visits as scheduled, well communicate with the investigators and complete the study as required by the study.

Exclusion Criteria:

1. Diagnosed as vascular immunoblastic t-cell lymphoma (AITL) or adult t-cell lymphoma/leukemia(ATLL);
2. Defined central nervous system (CNS) infiltration of lymphoma, including brain parenchyma, meningeal infringement or spinal cord compression;
3. Previous history of organ transplantation or allogeneic hematopoietic stem cell transplantation;
4. Patients who have active, known or suspected autoimmune diseases;
5. Patients who were previously treated with anti PD-1 antibody, anti PD-L1 antibody, anti PD-L2 antibody or anti CTLA-4 antibody (or any other antibodies acting on T cell co-stimulation or checkpoint pathway);
6. Complicated with other serious internal diseases, including but not limited to uncontrolled diabetes mellitus, active gastrointestinal ulcers, active hemorrhage, etc.;
7. Received treatment with other study drugs within 30 days before administration of the study drug or before 5 half-lives of other study drugs (whichever is shorter); or use of investigational medical device within 30 days;
8. Patients with active pulmonary tuberculosis; patients who previously had active pulmonary tuberculosis;
9. Any of the following is positive: hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), acquired immunodeficiency syndrome antibody (Anti-HIV) and anti-treponema pallidum antibody (TP-Ab);
10. Patients with complications requiring treatment with immunosuppressive drugs or systemic or local corticosteroids at the immunosuppressive doses;
11. Received treatment with other study drugs within 30 days before administration of the study drug or before 5 half-lives of other study drugs (whichever is shorter); or use of investigational medical device within 30 days;
12. Patients receiving any anti-infection vaccine (e.g. influenza vaccine, varicella vaccine etc.) within 4 weeks before enrollment;
13. Patients with symptomatic pleural, peritoneal and pericardial effusion;
14. Patients with drug abuse history or alcohol addiction history;
15. Uncontrollable or symptomatic dropsy of serous cavity, e.g. ascites, pleural effusion or pericardial effusion;
16. Lactating women;
17. Patients who had been previously treated with any other investigational drugs or participated in another clinical study within 30 days before enrollment;
18. Patients who are allergic to recombinant humanized antibody or any of its excipients;
19. Known allergies to recombinant humanized monoclonal antibody or any of its excipient components; A known history of severe allergic disease;
20. Patients who have insufficient communication, understanding and cooperation; or patients who have poor compliance and cannot guarantee to strictly follow the study protocol;
21. Subjects who are considered unsuitable for participating in this study for various reasons at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | up to 2 years
  To evaluate the efficacy of GB226 as defined by objective response rate in Chinese patients with recurrent or refractory PTCL

SECONDARY OUTCOMES:
Duration of response, DOR | up to 2 years
  To evaluate the duration of response (DOR) of GB226 in Chinese patients with recurrent or refractory PTCL
Overall survival, OS | up to 2 years
  To evaluate the duration from the first administration to death because of any reason in Chinese patients with recurrent or refractory PTCL
Progression-free survival, PFS | up to 2 years
  To evaluate the efficacy of GB226 as defined by progression-free survival, in Chinese patients with recurrent or refractory PTCL
Disease control rate (DCR) | up to 2 years
  To evaluate the efficacy of GB226 as defined by disease control rate, inChinese patients with recurrent or refractory PTCL
Time to response,TTR | up to 2 years
  To evaluate the efficacy of GB226 as defined by time to response in Chinese patients with recurrent or refractory PTCL
Antidrug antibody | up to 2 years
  To evaluate the immunogenicity of GB226 in Chinese patients with recurrent or refractory PTCL
Adverse Effect (AE) | up to 2 years
  To evaluate the adverse effect of GB226 in Chinese patients with recurrent or refractory PTCL

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Derived] Lou N, Yang M, Xie Z, Gao R, Zhang L, Tang L, Yao J, Han X, Shi Y. JAK3 A573V and JAK3 M511I mutations in peripheral T-cell lymphoma mediating resistance to anti-PD-1 therapy through the STAT3/PD-L1 pathway. J Immunother Cancer. 2025 Apr 8;13(4):e010783. doi: 10.1136/jitc-2024-010783. PMID 40199606
- [Derived] Shi Y, Wu J, Wang Z, Zhang L, Wang Z, Zhang M, Cen H, Peng Z, Li Y, Fan L, Guo Y, Ma L, Cui J, Gao Y, Yang H, Zhang H, Wang L, Zhang W, Zhang H, Xie L, Jiang M, Zhou H, Shuang Y, Su H, Ke X, Jin C, Du X, Du X, Liu L, Xi Y, Ge Z, Feng R, Zhang Y, Zhou S, Xie F, Wang Q. Efficacy and safety of geptanolimab (GB226) for relapsed or refractory peripheral T cell lymphoma: an open-label phase 2 study (Gxplore-002). J Hematol Oncol. 2021 Jan 12;14(1):12. doi: 10.1186/s13045-021-01033-1. PMID 33436023